CLINICAL TRIAL: NCT02870790
Title: Impact of the Rapid Expansion of Pre-exposure Prophylaxis (PrEP) on HIV Incidence, in a Setting With High HIV Testing and Antiretroviral Treatment Coverage, to Achieve the Virtual Elimination of HIV Transmission by 2020: a NSW HIV Strategy Implementation Project
Brief Title: Expanded PrEP Implementation in Communities in NSW
Acronym: EPIC-NSW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HEPP1511
Record Dates: First submitted 2016-08-14; First posted 2016-08-17 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: HIV; STI
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): A single open-label arm. All participants receive daily oral pill containing TDF/FTC
  Interventions: Drug: TDF/FTC

INTERVENTIONS:
Drug: TDF/FTC — one pill daily
  Other Names: Truvada; generic TDF/FTC

SUMMARY:
A new NSW Ministry of Health HIV Strategy released on 1 December 2015 aims for the virtual elimination of HIV transmission in NSW by 2020. Critical to the new strategy's success is the population-based, targeted roll-out of HIV PrEP. PrEP involves taking one pill daily of co-formulated tenofovir disoproxil fumarate (TDF)/ emtricitabine (FTC). This large-scale study aims for the rapid roll-out of TDF/FTC to individuals at high risk of HIV, who will comprise mostly gay and bisexual men (GBM) but will also include small numbers of heterosexuals, injecting drug users, and transgender men and women. The drug will be used according to existing NSW Ministry of Health Guidelines. By rapidly rolling out this new intervention over a 12 month period, and following participants for two years on treatments, a reduction of about 50% in new HIV diagnoses in NSW is expected.

The study aims to assess the incidence of HIV among PrEP study participants and measure the population-level impact of the rapid roll-out of PrEP on HIV diagnoses among GBM in NSW over a two-year period.

It will also evaluate the rate of PrEP uptake among high risk GBM in NSW, assess the incidence of STI (gonorrhoea, chlamydia and infectious syphilis) among people prescribed PrEP and measure the effect of the rapid roll-out of PrEP on the overall number of notifications of gonorrhoea, chlamydia and infectious syphilis in NSW, describe patterns of PrEP use and medication adherence, and monitor behavioural risk practices among PrEP users.

The main population group will be more than 3700 gay men at high risk of HIV infection. All procedures of this study are guided by the NSW Guidelines on PrEP.

Protocol Co-Chairs Professor David Cooper, Professor Andrew Grulich. Project Manager: Barbara Yeung

ELIGIBILITY:
Inclusion Criteria:

* HIV negative at enrolment, with a negative HIV test result documented within seven days of initiating PrEP
* At high and ongoing risk for acquiring HIV infection through sexual exposure (as defined by Behavioural Eligibility criteria presented in Appendix II and online Risk Assessment Questionnaire in Appendix III), OR previously a PrELUDE study participant
* Aged 18 years or over
* Live in NSW or ACT or visit NSW or ACT enough to attend clinics for follow-up assessments
* Willing and able to provide informed consent
* Medicare ineligible individuals may be enrolled if the clinical service is able to cover the costs of monitoring of the patient

Exclusion Criteria:

* HIV-1 infected or has symptoms consistent with acute viral infection (If HIV positive status is not confirmed by testing, delay starting PrEP for at least one month and reconfirm negative HIV-1 status).
* Having an estimated creatinine clearance (glomerular filtration rate [GFR]) <60ml/min
* Having or developing clinical symptoms suggestive of lactic acidosis or pronounced hepatotoxicity (including nausea, vomiting, unusual or unexpected stomach discomfort, and weakness)
* Concurrently taking a nephrotoxic agent (e.g., high-dose non-steroidal anti-inflammatory drugs / NSAIDs)
* Allergic to TDF and/or FTC (based on self-report or recorded)
* Concurrently taking prescribed products containing FTC or TDF including ATRIPLA®, COMPLERA®, EMTRIVA, STRIBILD®, VIREAD, TAF (tenofovir alafenamide), GENVOYA, DESCOVY; other drugs containing lamivudine; HEPSERA
* Factors or conditions that may compromise a participant's access to health services for follow-up (incarceration or planned relocation and potential absence from NSW or ACT).

Behavioural eligibility criteria as per NSW PrEP guidelines.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9733 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Incidence of HIV infection per 100 person years among study participants | 24 months of follow-up
Number of HIV diagnoses among gay and bisexual men notified to the NSW Ministry of Health. | 24 months of follow-up

SECONDARY OUTCOMES:
Incidence of STI (gonorrhoea, chlamydia and infectious syphilis) per 100 person years among study participants | 24 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David Cooper, MD, PhD, Study Chair — The Kirby Institute, UNSW Sydney; Andrew Grulich, MD, PhD, Study Chair — The Kirby Institute, UNSW Sydney
Locations (31):
- Australia (31):
  - Interchange General Practice, Canberra, Australian Capital Territory
  - Canberra Sexual Health Centre, Canberra, Australian Capital Territory
  - Albury Sexual Health Service, Albury, New South Wales
  - Fountain Street General Practice, Alexandria, New South Wales
  - Holdsworth House Byron Bay, Byron Bay, New South Wales
  - RPA Sexual Health, Camperdown, New South Wales
  - Coffs Harbour Sexual Health Clinic, Coffs Harbour, New South Wales
  - St Vincent's Hospital HIV, Immunology and Infectious Disease Unit, Darlinghurst, New South Wales
  - Dubbo Sexual Health, Dubbo, New South Wales
  - Dr Doong's Surgery, Enfield, New South Wales
  - Holden Street Gosford, Gosford, New South Wales
  - Illawarra Shoalhaven Sexual Health, Illawarra, New South Wales
  - Short Street Clinic, Kogarah, New South Wales
  - Lismore Sexual Health Clinic - Northen Rivers Area Health Service, Lismore, New South Wales
  - Liverpool Sexual Health Clinic, Liverpool, New South Wales
  - Hunter New England Sexual Health Services, Newcastle, New South Wales
  - St Leonards Medical Centre, North Sydney, New South Wales
  - Orange Sexual Health, Orange, New South Wales
  - Western Sydney Sexual Health Centre, Parramatta, New South Wales
  - Macleay Street Medical Practice, Potts Point, New South Wales
  - Crown Street Medical Centre, Surry Hills, New South Wales
  - The Albion Centre, Surry Hills, New South Wales
  - Kirketon Road Centre, Sydney, New South Wales
  - Sydney Sexual Health Centre, Sydney, New South Wales
  - East Sydney Doctors, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Taylor Square Private Clinic, Sydney, New South Wales
  - Clinic 16, Royal North Shore Hospital, Sydney, New South Wales
  - Nepean Sexual Health and HIV Clinic, Sydney, New South Wales
  - Brookong Centre Sexual Health Centre, Wagga Wagga, New South Wales
  - Green Square Health, Waterloo, New South Wales

REFERENCES:
- [Derived] Amin J, Vaccher S, Templeton DJ, Bavinton B, Jin F, Zablotska I, Matthews G, Ogilvie E, Yeung B, Ooi C, Dharan N, Baker DA, Read P, Guy R, Grulich AE. Low Prior Exposure and Incidence of Hepatitis C in Human Immunodeficiency Virus-Negative Gay and Bisexual Men Taking Preexposure Prophylaxis (PrEP): Findings From the Expanded PrEP Implementation in Communities-New South Wales Prospective Implementation Study. Clin Infect Dis. 2022 Oct 29;75(9):1497-1502. doi: 10.1093/cid/ciac231. PMID 35352102
- [Derived] Grulich AE, Jin F, Bavinton BR, Yeung B, Hammoud MA, Amin J, Cabrera G, Clackett S, Ogilvie E, Vaccher S, Vickers T, McNulty A, Smith DJ, Dharan NJ, Selvey C, Power C, Price K, Zablotska I, Baker DA, Bloch M, Brown K, Carmody CJ, Carr A, Chanisheff D, Doong N, Finlayson R, Lewis DA, Lusk J, Martin S, Ooi C, Read P, Ryder N, Smith D, Tuck Meng Soo C, Templeton DJ, Vlahakis E, Guy R; Expanded PrEP Implementation in Communities New South Wales (EPIC-NSW) research group. Long-term protection from HIV infection with oral HIV pre-exposure prophylaxis in gay and bisexual men: findings from the expanded and extended EPIC-NSW prospective implementation study. Lancet HIV. 2021 Aug;8(8):e486-e494. doi: 10.1016/S2352-3018(21)00074-6. Epub 2021 Jul 1. PMID 34217426
- [Derived] Grulich AE, Guy R, Amin J, Jin F, Selvey C, Holden J, Schmidt HA, Zablotska I, Price K, Whittaker B, Chant K, Cooper C, McGill S, Telfer B, Yeung B, Levitt G, Ogilvie EE, Dharan NJ, Hammoud MA, Vaccher S, Watchirs-Smith L, McNulty A, Smith DJ, Allen DM, Baker D, Bloch M, Bopage RI, Brown K, Carr A, Carmody CJ, Collins KL, Finlayson R, Foster R, Jackson EY, Lewis DA, Lusk J, O'Connor CC, Ryder N, Vlahakis E, Read P, Cooper DA; Expanded PrEP Implementation in Communities New South Wales (EPIC-NSW) research group. Population-level effectiveness of rapid, targeted, high-coverage roll-out of HIV pre-exposure prophylaxis in men who have sex with men: the EPIC-NSW prospective cohort study. Lancet HIV. 2018 Nov;5(11):e629-e637. doi: 10.1016/S2352-3018(18)30215-7. Epub 2018 Oct 17. PMID 30343026
- [Derived] Zablotska IB, Selvey C, Guy R, Price K, Holden J, Schmidt HM, McNulty A, Smith D, Jin F, Amin J, Cooper DA, Grulich AE; EPIC-NSW study group. Expanded HIV pre-exposure prophylaxis (PrEP) implementation in communities in New South Wales, Australia (EPIC-NSW): design of an open label, single arm implementation trial. BMC Public Health. 2018 Feb 2;18(1):210. doi: 10.1186/s12889-017-5018-9. PMID 29394918